CLINICAL TRIAL: NCT00064857
Title: Pycnogenol for the Treatment of Lymphedema of the Arm in Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001724-01 (NIH)
Record Dates: First submitted 2003-07-14; First posted 2003-07-16 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Lymphedema; Breast; Cancer
Keywords: lymphedema; breast; cancer; plant preparation; herbal preparation; pine bark extract
MeSH Terms: conditions — Lymphedema; Neoplasms | interventions — pycnogenols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pycnogenol

SUMMARY:
The goal of this study is to evaluate the effectiveness of a standardized botanical extract of Pycnogenol as a treatment for stable arm lymphedema in breast cancer survivors.

DETAILED DESCRIPTION:
Lymphedema of the arm affects the function and self-image of approximately 600,000 of the 2 million breast cancer survivors in the United States. Chronic lymphedema can lead to recurrent infections and permanent swelling, in some cases impairing function. Although various methods of massage and the use of non-elastic compression "sleeves" have been shown to decrease the severity of lymphedema, these methods of physical therapy are limited in terms of patient acceptance, compliance, and by the availability of trained therapists. There is presently no pharmacologic treatment that has proven effective in treating or preventing the development of lymphedema in women treated for breast cancer. This is a double-blind, placebo-controlled trial of an extract of the bark of the French maritime pine tree (Pycnogenol(r)) as a treatment for arm lymphedema in breast cancer survivors. Pycnogenol(r) is widely used in Europe for lymphedema of the leg and varicose veins, and is thought to act by several mechanisms including vascular permeability and vascular constriction. The development of such a therapeutic approach would therefore constitute a major breakthrough in the treatment of this common symptom of breast cancer lymphedema. Bioelectric impedance is a painless, quick, and easily-performed method of estimating the extracellular and total water volume of the body or segment, such as the arm. We will compare the correlation of both a single- and a multiple-frequency bioelectric impedance instrument in measuring change in arm volume to a standard assessment using water displacement. We expect that bioelectric impedance will prove faster and more sensitive to changes in extracellular water (lymphedema) than the water displacement method. We also propose to use a small oral dose of midazolam and single blood sampling to screen for effects of Pycnogenol(r) on the activity of the common drug metabolizing enzyme CYP3A4. For those subjects who are already receiving digoxin, we will use digoxin urine excretion to screen for effects of the botanical upon the activity of P-glycoprotein. Finally, we will continue the evaluation of a new questionnaire of lymphedema symptoms presently being tested as a tool for assessing the severity and improvement of symptoms with treatment. In summary, the successful completion of this research can be expected to provide an alternative therapy and new instruments for treating and measuring lymphedema.

ELIGIBILITY:
Inclusion criteria:

* Unilateral (ipsilateral to breast cancer resection side) lymphedema of the upper extremity.
* Extravascular water ration of > 1.07/1 between affected vs. normal arm using multiple frequency bioelectric impedence
* Patient is > 2months from last surgical or radiation treatment to the affected axilla
* Renal and hepatic function:

Creatinine clearance > 50ml/min, total bili <2 mg/dl, transaminases <1.5 x ULN

* Patient not pregnant or breastfeeding. Use of barrier contraception if sexually active.
* ECOG performance of 0-2
* Patient not allergic to pycnogenol

Exclusion criteria:

* Patients treated with their first course of chemotherapy or radiation
* Chemotherapy or radiation to axillary lymph node will exclude patients for 8 weeks following treatment
* Patients with more than one episode of arm cellulitis, venous clot, or woody fibrosis of the affected arm. Antibiotics used to treat cellulitis must be completed at least 4 weeks prior to initial screening
* Patients with a defibrillator Midazolam study only: Patients requiring or benefiting from supplemental oxygen, patients allergic to cherries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2003-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Cleary, M.B.B.S., Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center and School of Pharmacy, Madison, Wisconsin, United States